CLINICAL TRIAL: NCT06233110
Title: Phase I Trial of Ruxolitinib Plus Fostamatinib for the Treatment of Steroid Refractory Chronic Graft Versus Host Disease
Brief Title: Ruxolitinib Plus Fostamatinib for Steroid Refractory cGvHD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stefanie Sarantopoulos, MD, PhD. (Other)
Collaborators: Incyte Corporation (Industry); Rigel Pharmaceuticals (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Stefanie Sarantopoulos, MD, PhD., Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00113327
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — fostamatinib; ruxolitinib

STUDY DESIGN:
Intervention Model Description: Initial dose escalation cohort:
  Subjects enrolled in the initial dose escalation cohort will begin combination therapy with ruxolitinib 10mg twice daily and fostamatinib 100mg daily (dose level 1). As dictated by the 3+3 design, the dose of fostamatinib for subsequent patients will be 150mg daily (dose level 2) or 100mg twice daily (dose level 3). A dose level 0 of fostamatinib at 50mg daily will be evaluated if the frequency of dose-limiting toxicities at dose level 1 prevents the selection of a biologically optimal dose.
  Safety expansion cohort:
  Fostamatinib will be given at one of two identified candidate doses from the dose escalation cohort. Subjects will be randomized to one of these two doses. A total of 12 subjects will be accrued for each candidate dose level, including those who received the candidate doses in the dose escalation phase. Subjects will receive ruxolitinib at a dose of 10mg twice daily.
Who Masked: Participant
Masking Description: In the subsequent safety expansion cohort, patients will be randomized to one of the two selected candidate doses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose escalation phase: Dose level 0 (Experimental): Fostamatinib at dose level 0 (dose of 50mg QAM) in combination with standard of care ruxolitinib 10mg BID
  Interventions: Drug: Fostamatinib; Drug: Ruxolitinib
- Dose escalation phase: Dose level 1 (Experimental): Fostamatinib at dose level 1 (dose of 100mg QAM) in combination with standard of care ruxolitinib 10mg BID
  Interventions: Drug: Fostamatinib; Drug: Ruxolitinib
- Dose escalation phase: Dose level 2 (Experimental): Fostamatinib at dose level 2 (dose of 150mg QAM) in combination with standard of care ruxolitinib 10mg BID
  Interventions: Drug: Fostamatinib; Drug: Ruxolitinib
- Dose escalation phase: Dose level 3 (Experimental): Fostamatinib at dose level 3 (dose of 100mg BID) in combination with standard of care ruxolitinib 10mg BID
  Interventions: Drug: Fostamatinib; Drug: Ruxolitinib
- Candidate Dose #1 (Experimental): In the safety expansion cohort, subjects will be randomized to one of two candidate doses of fostamatinib (identified from the dose escalation phase) in combination with ruxolitinib 10mg BID.
  Interventions: Drug: Fostamatinib; Drug: Ruxolitinib
- Candidate Dose #2 (Experimental): In the safety expansion cohort, subjects will be randomized to one of two candidate doses of fostamatinib (identified from the dose escalation phase) in combination with ruxolitinib 10mg BID.
  Interventions: Drug: Fostamatinib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Fostamatinib — Fostamatinib will be administered as part of the initial dose escalation cohort and then two candidate doses will be identified to be administered for the safety expansion cohort.
Drug: Ruxolitinib — Ruxolitinib 10mg BID will be administered in combination with Fostamatinib in each of the study arms.

SUMMARY:
This is an open-label phase I study of fostamatinib in combination with ruxolitinib for the treatment of chronic GvHD with a suboptimal response to corticosteroids. The primary objective is to identify a minimum safe and biologically effective dose of fostamatinib when combined with standard of care ruxolitinib for the treatment of steroid refractory and steroid dependent cGVHD. The secondary objective is to estimate the efficacy of the combination of ruxolitinib and fostamatinib for the treatment of steroid refractory and steroid dependent cGVHD.

The target enrollment is 24-30 subjects. The study will begin with an initial dose escalation cohort employing a modified 3+3 design to investigate up to three doses of fostamatinib. Using safety, efficacy, pharmacodynamic (PD), and pharmacokinetic data (PK), an interim assessment will be performed to determine two candidate doses of the biologically optimal dose to investigate further. A safety expansion cohort will be opened to backfill these two candidate doses up to a total 12 patients per dose, including those in the dose escalation cohort who received the candidate doses. Patients will then be randomized to one of these two candidate doses in the expansion. If there is an imbalance in the two expansion cohorts, the remaining patient slots after 1:1 randomization will be sequentially backfilled to a total of 12 patients per cohort. A final analysis of safety, efficacy, and PK/PD data in patients who received the two candidate doses will be conducted to determine a minimum safety and biologically effective dose, which will be the recommended phase II dose (RP2D).

The primary hypothesis is that Fostamatinib combined with ruxolitinib is a safe therapy for and has synergistic activity in cGvHD. The recommended phase II dose will be determined by the study investigators in collaboration with the sponsors. The decision to select the recommended phase II dose will occur only after all patients in the part 1 have completed at least 28 days of therapy. The decision will be based on the valuation of all relevant, available data, and not solely on dose-limiting toxicities.

ELIGIBILITY:
Inclusion Criteria

1. Patient is able and willing to provide written informed consent prior to any study related screening procedures are performed.
2. Age ≥ 18 years old at the time of informed consent
3. Have undergone allogeneic hematopoietic cell transplantation (HCT) from any donor source (matched unrelated donor, sibling, haploidentical) using bone marrow, peripheral blood, or cord blood stem cells.
4. Adequate bone marrow function defined as:

   4.1 Absolute neutrophil count (ANC) ≥ 750 /mm3 4.2 Platelet count ≥ 40,000 /mm3 4.3 Hemoglobin ≥ 8.0 g/dL without transfusion support Note: Use of growth factor supplementation (myeloid, erythroid or megakaryocytic) is permitted to meet eligibility criteria.
5. Patients with clinically diagnosed cGvHD staging of mild to severe according to NIH Consensus Criteria4 prior to Cycle 1 Day 1 and with confirmed steroid refractoriness or steroid dependence irrespective of the concomitant use of a calcineurin inhibitor, as follows:

   5.1 Disease progression after administration of a minimum dose of 1.0 mg/kg/day or equivalent for at least 1 week at any time following diagnosis of cGvHD OR 5.2 Disease persistence despite continued treatment with prednisone > 0.5mg/kg/d or equivalent for at least 4 weeks OR 5.3 Increase to prednisone > 0.25 mg/kg/d after 1 unsuccessful attempt to taper the dose.

   5.4 Recurrence of chronic GVHD after attaining a complete response 5.5 Progression of chronic GVHD after attaining a partial response
6. Patient has Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Exclusion Criteria

1. Prior or ongoing treatment with ruxolitinib for treatment of cGvHD for longer than 3 weeks prior to anticipated C1D1.
2. Prior treatment with fostamatinib or another SYK inhibitor for the treatment of acute or chronic GVHD. Prior use of fostamatinib for conditions other than GVHD is permitted.
3. Ongoing systemic therapy for cGvHD other than corticosteroids, calcineurin inhibitor, or mycophenolate mofetil, aside from fewer than 3 weeks of ruxolitinib. Prior ruxolitinib use for the indication of acute GVHD is permitted.
4. Patients with relapsed primary malignancy, or who have been treated for relapse after the allogeneic HCT was performed
5. SR-cGvHD occurring after a non-scheduled donor lymphocyte infusion (DLI) administered for pre-emptive treatment of malignancy recurrence. Patients who have received a scheduled DLI as part of their transplant procedure and not for management of malignancy relapse are eligible.
6. History of progressive multifocal leuko-encephalopathy (PML)
7. Active uncontrolled bacterial, fungal, parasitic, or viral infection. Infections are considered controlled if appropriate therapy has been instituted and, at the time of screening, no signs of infection progression are present.
8. Clinical evidence of active and clinically significant viral disease including HIV, CMV, HHV-6, HBV, HCV, or BK virus.
9. Patients on mechanical ventilation or have a resting O2 saturation < 90% by pulse oximetry
10. Clinically significant and uncontrolled cardiovascular disease, including unstable angina, acute myocardial infarction, or stroke within 3 months, or NYHA Class III or IV congestive heart failure.
11. Uncontrolled hypertension with systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg.
12. Creatinine clearance by Cockcroft-Gault of < 15 mL/min and not on dialysis
13. Total bilirubin > 3 times ULN, ALT > 5 times ULN, or AST > 5 times ULN
14. QTc ≥ 470 ms as calculated by the Fridericia Formula
15. Active pregnancy or breast feeding, or currently seeking active pregnancy
16. Any patient who, in the opinion of the investigator, may not be able to comply with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Minimum safe and biologically effective dose | 6 months
  Minimum safe and biologically effective dose will be determined by dose limiting toxicities and overall response rate of the combination regimen, as well as pharmacokinetic and pharmacodynamic markers of fostamatinib (if available)

SECONDARY OUTCOMES:
Overall response rate | 6 months
  Overall response rate, as defined by achievement of a complete response (CR) or partial response (PR), using the 2014 NIH Consensus criterion, during the first 6 months of therapy.
Duration of Response | 1 year
  The length of time that a patient's response to treatment lasts.
1-year cGvHD-free survival | 1 year
  The cGVHD-free survival is a composite endpoint that measures survival free from the diagnosis of chronic GVHD at any stage. cGvHD activity assessment includes medical history, physical exam, and laboratory studies per the 2014 NIH Consensus Response Criteria.
Overall survival | 1 year
  The length of time that a patient lives following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chenyu Lin, MD, Principal Investigator — Duke Health
Locations (1):
- Duke, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No